CLINICAL TRIAL: NCT02397473
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients With Episodic Cluster Headache
Brief Title: A Study Of Galcanezumab In Participants With Episodic Cluster Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15780; I5Q-MC-CGAL (Other: Eli Lilly and Company); 2015-000149-22 (EudraCT Number)
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Episodic Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Galcanezumab 300mg (Experimental): Galcanezumab 300mg administered subcutaneously (SC) every 30 days during an 8 week treatment period.
  Interventions: Drug: Galcanezumab
- Placebo (Placebo Comparator): Placebo administered SC every 30 days during an 8 week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742
  Arms: Galcanezumab 300mg
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of the study drug known as Galcanezumab in participants with episodic cluster headaches.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cluster headache as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta guidelines with a history of episodic cluster headache with at least two cluster periods lasting from 7 days to 1 year (when untreated) and separated by pain-free remission periods of >=1 month.
* Participants are able to distinguish cluster headache attacks from other headaches.

Exclusion Criteria:

* Current enrollment in or discontinuation within the last 30 days from, a clinical trial involving any investigational drug or device.
* Current use or any prior exposure to any calcitonin-gene-related peptide (CGRP) antibody, any antibody to the CGRP receptor, or antibody to nerve growth factor (NGF).
* Are taking indomethacin and/or are suspected of having another distinct trigeminal autonomic cephalalgia.
* A history of migraine variants that could implicate or could be confused with ischemia.
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins.
* A history or presence of other medical illness that indicates a medical problem that would preclude study participation.
* Evidence of significant active or unstable psychiatric disease, in the opinion of the investigator.
* Women who are pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (46):
- United States (17):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford University Hospital, Palo Alto, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Colorado Neurological Institute, Englewood, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - St. Anthony's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Michigan Head, Pain, and Neurological Institute, Ann Arbor, Michigan
  - ClinVest, Springfield, Missouri
  - Dent Neurological Institute, Amherst, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Northwest Clinical Research Center, Bellevue, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Liège
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Glostrup Municipality, Denmark
- Finland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jyväskylä
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Turku
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Paris
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
- Germany (4):
  - Uniklinikum Essen AöR, Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Hamburg
  - Migräne- und Kopfschmerzklinik GmbH & Co. KG, Königstein
  - Klinikum der Universität München Campus Großhadern, München
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Greece
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pavia
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Valencia
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Hull
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Liverpool
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., London

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Jensen RH, Tassorelli C, Myers Oakes TM, Bardos JN, Zhou C, Dong Y, Aurora SK, Martinez JM. Baseline demographics and disease characteristics of patients with episodic or chronic cluster headache: data from two phase 3 randomized clinical trials in Europe and North America. Front Neurol. 2023 Dec 15;14:1293163. doi: 10.3389/fneur.2023.1293163. eCollection 2023. PMID 38162453
- [Derived] Andrews JS, Kudrow D, Rettiganti M, Oakes T, Bardos JN, Wenzel R, Kuruppu DK, Gaul C, Martinez JM. Impact of Galcanezumab on Total Pain Burden: A Post Hoc Analysis of a Phase 3, Randomized, Double-Blind, Placebo-Controlled Study in Patients with Episodic Cluster Headache. J Pain Res. 2021 Jul 8;14:2059-2070. doi: 10.2147/JPR.S305066. eCollection 2021. PMID 34267550
- [Derived] Goadsby PJ, Dodick DW, Leone M, Bardos JN, Oakes TM, Millen BA, Zhou C, Dowsett SA, Aurora SK, Ahn AH, Yang JY, Conley RR, Martinez JM. Trial of Galcanezumab in Prevention of Episodic Cluster Headache. N Engl J Med. 2019 Jul 11;381(2):132-141. doi: 10.1056/NEJMoa1813440. PMID 31291515
- See also: Click here for more information about this study: A Study of LY2951742 in Participants With Episodic Cluster Headache — https://www.lillytrialguide.com/en-US/studies/episodic-cluster-headache/CGAL

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo once a month for 2 months by subcutaneous (SC) injection.
  Participants did not receive any intervention during post treatment follow-up phase.
- Galcanezumab 300mg: Participants received Galcanezumab 300mg once a month for two months by subcutaneous (SC) injection.
  Participants did not receive any intervention during post treatment follow-up phase.
Period: Treatment Phase
Arm/Group | Placebo | Galcanezumab 300mg
Started | 57 | 52
Received at Least One Dose of Study Drug | 57 | 49
Completed | 45 | 45
Not Completed | 12 | 7
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 8 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation(did not receive drug) | 0 | 3
Period: Post Treatment Follow-up Phase
Arm/Group | Placebo | Galcanezumab 300mg
Started | 50 (Participants who discontinued treatment period had an option to enter post treatment phase.) | 47
Completed | 47 | 45
Not Completed | 3 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo once a month for 2 months by SC injection.
  Participants did not receive any intervention during post treatment follow-up phase.
- Galcanezumab 300mg: Participants received Galcanezumab 300mg once a month for two months by SC injection.
  Participants did not receive any intervention during post treatment follow-up phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | Galcanezumab 300mg | Total
Number analyzed (Participants) | 57 | 49 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.40 (11.32) | 47.49 (10.74) | 46.37 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 47 | 41 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 45 | 41 | 86
  Unknown or Not Reported | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 47 | 43 | 90
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 1 | 2 | 3
  Canada | 1 | 1 | 2
  Netherlands | 1 | 2 | 3
  Belgium | 4 | 4 | 8
  United States | 18 | 16 | 34
  Finland | 2 | 1 | 3
  Denmark | 2 | 1 | 3
  Italy | 11 | 9 | 20
  United Kingdom | 1 | 1 | 2
  France | 5 | 4 | 9
  Germany | 4 | 2 | 6
  Spain | 7 | 6 | 13
Weekly Cluster Headache Attacks [Mean (Standard Deviation); unit: Cluster Headache Attacks per week] | 17.30 (10.05) | 17.82 (10.12) | 17.54 (10.04)
Lifetime suicidal ideation prior to screening [Count of Participants; unit: Participants] | 5 | 9 | 14
Lifetime suicidal behavior prior to screening [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in Number of Weekly Cluster Headache Attacks
Description: Number of cluster headache attacks was recorded daily by study participants in their ePRO Diary. Overall mean change from baseline is derived from the average of weeks 1 to 3 from mixed model repeated measures (MMRM) analysis. Least Square (LS) means were calculated using MMRM model with treatment, sex, pooled investigative site, week, baseline, and treatment by week as fixed effects.
Time Frame: Baseline, Week 1 through Week 3
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Cluster Headache Attacks per Week
Groups:
- Placebo: Participants received placebo once a month for two months by SC injection.
  Participants did not receive any intervention during post treatment follow-up phase.
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 57 | 49
Cluster Headache Attacks per Week | -5.22 (1.33) | -8.69 (1.42)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300mg; Test type: Superiority; p = 0.036, Mixed Models Analysis; LSMean Difference = -3.47, 95% CI 2-sided [-6.72 to -0.23], Standard Error of Mean 1.63

2. Secondary Outcome: Percentage of Participants With 50% or Greater Reduction From Baseline in the Weekly Number of Cluster Headache Attacks
Description: Number of cluster headache attacks was recorded daily by study participants in their ePRO Diary. Percentage of participants with 50% or greater reduction from baseline at week 3 was analyzed using Koch's nonparametric randomization-based analysis of covariance method. This method adjusted for pooled investigative site by including it as a stratification variable. It also adjusted for sex and baseline value.
Time Frame: Baseline, Week 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 57 | 49
percentage of participants | 52.63 | 71.43
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300mg; Test type: Superiority; p = 0.046, ANCOVA; Koch's nonparametric randomization-based ANCOVA

3. Secondary Outcome: Overall Mean Change From Baseline in Number of Weekly Cluster Headache Attacks
Description: Number of cluster headache attacks was recorded daily by study participants in their ePRO Diary. Overall mean change from baseline is derived from the average of weeks 1 to 8 from MMRM analysis. Least Square (LS) means were calculated using MMRM model with treatment, sex, pooled investigative site, week, baseline, and treatment by week as fixed effects.
Time Frame: Baseline, Week 1 through Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Cluster Headache Attacks per Week
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 57 | 49
Cluster Headache Attacks per Week | -9.97 (0.95) | -10.80 (1.00)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300mg; Test type: Superiority; p = 0.493, Mixed Models Analysis; LSMean Difference = -0.83, 95% CI 2-sided [-3.23 to 1.57], Standard Error of Mean 1.20

4. Secondary Outcome: Percentage of Participants Reporting a Score of 1 or 2 on the Patient Global Impression of Improvement (PGI-I)
Description: PGI-I requests participants to mark the box that best describes their cluster headache condition since they started taking the medicine. The options in the displayed boxes are represented on a 7-point scale, with 1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, and 7 = very much worse. Percentage of participants were derived with a generalized linear mixed model repeated measures method with treatment, sex, baseline cluster headache attack category, month, and treatment by month as fixed effects.
Time Frame: Week 4
Population: All randomized participants who received at least one dose of study drug and had PGI-I measurement at week4.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 49 | 44
percentage of participants | 46.4 | 72.5
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300mg; Test type: Superiority; p = 0.016, Mixed Models Analysis; Odds Ratio (OR) = 3.046, 95% CI 2-sided [1.242 to 7.469]

5. Secondary Outcome: Percentage of Participants Reporting a Score of 1 or 2 on the Patient Global Impression of Improvement (PGI-I)
Description: as for outcome 4
Time Frame: Week 8
Population: All randomized participants who received at least one dose of study drug and had PGI-I measurement at week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 40 | 38
percentage of participants | 66.1 | 71.9
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300mg; Test type: Superiority; p = 0.575, Mixed Models Analysis; Odds Ratio (OR) = 1.312, 95% CI 2-sided [.502 to 3.426]

6. Secondary Outcome: Percentage of Participants With 50% or Greater Reduction From Baseline in Number of Weekly Cluster Headache Attacks
Description: Number of cluster headache attacks was recorded daily by study participants in their ePRO Diary. Mean percentage of participants is derived from the average of weeks 1 to 8 from generalized linear mixed model repeated measures method with treatment, sex, week, treatment by week, and baseline as fixed effects.
Time Frame: Baseline, Week 1 through Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 57 | 49
percentage of participants | 70.4 | 69.6
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300mg; Test type: Superiority; p = 0.910, Mixed Models Analysis; Pseudo-likelihood-based repeated measures; Odds Ratio (OR) = .965, 95% CI 2-sided [.512 to 1.819]

7. Secondary Outcome: Percentage of Participants With 30% or Greater Reduction From Baseline in Number of Weekly Cluster Headache Attacks
Description: Number of cluster headache attacks was recorded daily by study participants in their ePRO Diary. Mean percentage of participants is derived from the average of weeks 1 to 8 from generalized linear mixed model repeated measures with treatment, sex, week, treatment by week and baseline as fixed effects.
Time Frame: Baseline, Week 1 through Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 57 | 49
percentage of participants | 78.9 | 77.7
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 300mg; Test type: Superiority; p = 0.841, Mixed Models Analysis; Pseudolikelihood-based repeated measures model; Odds Ratio (OR) = 0.929, 95% CI 2-sided [0.449 to 1.923]

8. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Time Frame: Week 4
Population: All randomized participants who received at least one dose of study drug and had measurable PK samples.
Measure: Mean (Standard Deviation); unit: Nanogram per Milliliter (ng/mL)
Arm/Group | Galcanezumab 300mg
Number analyzed (Participants) | 45
Nanogram per Milliliter (ng/mL) | 20200 (6880)

9. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Time Frame: Week 8
Population: All randomized participants who received at least one dose of study drug and had measurable PK samples.
Measure: Mean (Standard Deviation); unit: Nanogram per Milliliter (ng/mL)
Arm/Group | Galcanezumab 300mg
Number analyzed (Participants) | 45
Nanogram per Milliliter (ng/mL) | 26400 (11200)

10. Secondary Outcome: Percentage of Participants Developing Anti-Drug Antibodies (ADA) to Galcanezumab
Description: Treatment emergent (TE) ADA evaluable participant is considered to be TE ADA+ if the subject has at least one post-baseline titer that is a 4-fold or greater increase in titer from baseline measurement. If baseline result is ADA Not Present, then the participant is TE ADA+ if there is at least one post-baseline result of ADA present with titer >= 1: 20.
Time Frame: Baseline through Week 8
Population: All randomized participants who received at least one dose of study drug and had non-missing baseline ADA result, and at least one non-missing post baseline ADA result.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 53 | 48
percentage of participants | 0 | 0

11. Secondary Outcome: Percentage of Participants With Suicidal Ideation Assessed by Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred. Some questions are binary responses (yes/no) and some are on a scale of 1 (low severity) to 5 (high severity). Suicidal ideation: a "yes" answer to any of 5 suicidal ideation questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods without intent to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent.
Time Frame: Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug and had at least one post baseline C-SSRS assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 54 | 49
percentage of participants | 0 | 0

12. Secondary Outcome: Percentage of Participants With Suicidal Behaviors Assessed by Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred. Some questions are binary responses (yes/no) and some are on a scale of 1 (low severity) to 5 (high severity). Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide.
Time Frame: Month 1 through Month 6
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 300mg
Number analyzed (Participants) | 54 | 49
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Groups:
- Placebo - Treatment Phase: Participants received placebo once a month for two months by SC injection.
- Galcanezumab 300mg - Treatment Phase: Participants received Galcanezumab 300mg once a month for two months by SC injection.
- Placebo - Post Treatment Phase; Galcanezumab 300mg - Post Treatment Phase: Participants didn't receive any intervention.
Arm/Group | Placebo - Treatment Phase | Galcanezumab 300mg - Treatment Phase | Placebo - Post Treatment Phase | Galcanezumab 300mg - Post Treatment Phase
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/49 | 0/50 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/49 | 2/50 | 0/47
Other Adverse Events (participants affected / at risk) | 4/57 | 7/49 | 3/50 | 1/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Treatment Phase (N=57) | Galcanezumab 300mg - Treatment Phase (N=49) | Placebo - Post Treatment Phase (N=50) | Galcanezumab 300mg - Post Treatment Phase (N=47)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Treatment Phase (N=57) | Galcanezumab 300mg - Treatment Phase (N=49) | Placebo - Post Treatment Phase (N=50) | Galcanezumab 300mg - Post Treatment Phase (N=47)
Injection site pain (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information provided to Investigator &/or Institution by Lilly or Lilly-designated representatives, or generated by Investigator &/or institution in connection with Study, will be kept in confidence and not used for any purpose not expressly provided in the Agreement for at least 5 years after termination or conclusion of Study, except to the extent that Lilly gives Investigator &/or Institution written permission or particular information is required by laws or regulations to be disclosed.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT02397473/SAP_000.pdf
  • Study Protocol (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT02397473/Prot_001.pdf